CLINICAL TRIAL: NCT02391389
Title: VentFirst Pilot: Ventilating Preterm Infants During Delayed Cord Clamping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Karen Fairchild, MD, Professor of Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17444
Record Dates: First submitted 2014-12-08; First posted 2015-03-18 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Infant, Premature, Diseases
Keywords: preterm infant
MeSH Terms: conditions — Infant, Premature, Diseases; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP or PPV during DCC (Experimental): Infant will receive CPAP or PPV from 30 to 90 seconds after birth while attached to the placenta, and then the umbilical cord will be cut at 90 seconds
  Interventions: Procedure: CPAP or PPV during DCC

INTERVENTIONS:
Procedure: CPAP or PPV during DCC — CPAP or PPV is provided during delayed cord clamping

SUMMARY:
Delayed clamping of the umbilical cord (DCC) has been shown to have some benefits for preterm infants. Initiation of breathing before cord clamping is also thought to be beneficial. Since some preterm infants do not breathe well on their own immediately after birth, assisting ventilation during delayed cord clamping might have additional benefit beyond DCC alone. "VentFirst Pilot" will assess feasibility and safety of assisting ventilation of preterm infants during 90 seconds of DCC which is essential before proceeding to a randomized clinical trial.

DETAILED DESCRIPTION:
Mothers expected to deliver an infant at 24-32 completed weeks' gestation will be approached for consent. When the infant is delivered, members of the neonatology team will be at the mother's side and will provide initial steps of resuscitation (position, suction, stimulate) per guidelines of the Neonatology Resuscitation Program (NRP). At 30 seconds after birth, the infant will receive continuous positive airway pressure (CPAP) if breathing well, or positive pressure ventilation (PPV) if not breathing well. At 90 seconds, the umbilical cord will be cut and the remainder of the resuscitation and stabilization will be carried out in the usual location.

ELIGIBILITY:
Inclusion Criteria:

- 24 0/7 to 32 6/7 weeks gestation at birth

Exclusion Criteria:

* major congenital anomalies
* monochorionic twins
* twin-twin transfusion syndrome
* hydrops fetalis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of deliveries in which providing ventilatory assistance during delayed cord clamping is achieved | 90 seconds after birth
  Assess the feasibility of the neonatology team performing initial resuscitation and providing ventilation during 90 seconds of delayed cord clamping

SECONDARY OUTCOMES:
Number of unanticipated complications of neonatal resuscitation during delayed cord clamping (neonatal temperature, hematocrit, bilirubin,maternal infection, and other clinical variables) | 7 days from birth
  Assess neonatal temperature, hematocrit, bilirubin,maternal infection, and other clinical variables

CONTACTS AND LOCATIONS:
Overall Officials: Karen D Fairchild, MD, Principal Investigator — University of Virginia SOM
Locations (1):
- University of Virginia School of Medicine, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Winter J, Kattwinkel J, Chisholm C, Blackman A, Wilson S, Fairchild K. Ventilation of Preterm Infants during Delayed Cord Clamping (VentFirst): A Pilot Study of Feasibility and Safety. Am J Perinatol. 2017 Jan;34(2):111-116. doi: 10.1055/s-0036-1584521. Epub 2016 Jun 15. PMID 27305177